# **CATSTAT-HF**



## Official Title of the study:

Serum Catestatin Expression and Cardiometabolic Parameters in Patients With

Congestive Heart Failure (CATSTAT-HF)

**NCT** number:

NCT03389386

### Date of the document:

April 15th 2019

## **Study organizations:**

University of Split School of Medicine University Hospital of Split







## STUDY ANALYSIS PLAN (SAP)

All data analyses will be performed by using IBM SPSS Statistics for Windows, version 23.0 (IBM Corp., Armonk, NY, USA) and/or Graphpad Prism 7 for Windows (GraphPad Software, Inc., La Jolla, CA, USA). All p-values in this study will be 2-tailed and results that reach p<0.05 will be considered statistically significant.

#### **GENERAL STATISTICAL ANALYSES:**

- 1. Descriptive analyses will provide data on particular categories of interest by using frequencies and percentages. Baseline sociodemographic, anthropometric and comorbidity burden data will be provided for each particular category.
- 2. A standard **Pearson's chi-squared test** will be used to determine statistical differences in categorical variables between the two groups of interest congestive heart failure-CHF patients vs. healthy volunteer controls and other potential subgroups of interest.
- 3. The unpaired **t-test** or **Mann-Whitney U-test**, based on the data distribution normality, will be used to determine statistical differences in continuous parameters between the two groups of interest *CHF patients vs. healthy volunteer controls* and other potential subgroups of interest, as needed. Continuous variables will be expressed as mean ± standard deviation (SD) or median ± interquartile range (IQR), based on the normality distribution.
- 4. **Bivariate Pearson correlation test (r)** is a parametric test that will be used to determine the significance of linear correlation between two continuous variables of interest (X, Y). In the determination of statistical correlation between continuous variables, a **multiple linear regression**, adjusted for confounders, will be used.

#### **SPECIFIC STATISTICAL ANALYSES:**

1. The analysis of variance (ANOVA) with post-hoc Tukey HSD test will be used to

determine statistical differences in continuous parameters among the three or more

subgroups of patients with CHF.

2. Receiver operating characteristics (ROC) curve analysis will be used to ascertain the

diagnostic sensitivity and specificity as well as corresponding cut-off values of serum

catestatin in determining heart failure (HF) degree and severity, e.g. rule out, rule in.

3. All multivariable regression analyses will be, at minimum, adjusted for age, sex, estimated

glomerular filtration rate (eGFR), and body mass index (BMI). Other important factors such as

medication intake and other potential confounding factors will be used in determining odds

ratios (OR) for the disease status (congestive heart failure). Adjusted ORs, statistical

significance (p) and 95% confidence intervals (95% CI) will be provided for independent

predictors.

Study statistical plan is provided and revised on

April 15th 2019 by

Josip A. Borovac, MD, BSc

josip.borovac@me.com

12-